CLINICAL TRIAL: NCT00789464
Title: H-23187: Probiotic Prophylaxis Against Recurrent Pediatric Urinary Tract Infection
Brief Title: Probiotics for Girls With Recurring Urinary Tract Infections
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn by PI
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Roth, Professor, TCH Urology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-23187
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Urinary Tract Infection; Probiotics; Dietary Supplements; Bacteriuria
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Other): Probiotics drops plus placebo elixir
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938
- ARM B (Other): TMP/SMZ elixir plus placebo drops
  Interventions: Drug: trimethoprim/sulfamethoxazole

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — DSM 17938 drops (10^8 cfu/dose of 5 drops) + placebo elixir once daily for 1 year.
  Arms: ARM A
Drug: trimethoprim/sulfamethoxazole — Trimethoprim/sulfamethoxazole elixir (TMP/SMZ) (2 mg/kg), a standardized oral antibiotic prophylaxis, plus placebo capsule once daily for 1 year.
  Other Names: TMP/SMZ, Bactrim, Septra
  Arms: ARM B

SUMMARY:
Probiotics are dietary supplements containing potentially beneficial bacterial strains such as Lactobacillus. The safety of oral administration of probiotics has been demonstrated in hundreds of studies using adults over the last 30 years. Very few studies have been conducted with children. UTI in girls occur when virulent bacteria migrate from the rectum and colonize the vagina and peri-urethral mucosa, thus gaining access to the bladder.

This study will randomize girls to ARM A (probiotics + placebo) and ARM B (antibiotics + placebo) to determine if UTIs are decreased when the probiotics are given.

ELIGIBILITY:
Inclusion Criteria:

* Girls age 1 through age 17 years of age
* Must have had at least 3 symptomatic UTI, uncomplicated or complicated, in the year preceding study inclusion or already using any form of prophylaxis to prevent recurrences of UTI
* Must have had at least 3 symptomatic urinary tract infections in the year before the start of the prophylaxis.

Exclusion Criteria:

* Breastfeeding
* Pregnancy
* Prior adverse reaction to sulfa drugs or sulfamethoxazole/trimethoprim
* Known immunosuppression i.e., transplant recipients or children with congenital immunodeficiencies
* Poorly controlled diabetes
* Untreated HIV infection
* Use of high dose corticosteroids for autoimmune diseases or post-organ transplantation. Inhaled corticosteroids or oral steroids for asthma are allowed.
* Malnutrition
* Patients with a history of sulfamethoxazole/trimethoprim-resistant UTI will be excluded from the study
* Patients with renal insufficiency, liver insufficiency, or cardiopulmonary disease requiring medication will be excluded from the study
* Patients with known anemia will be excluded from the study
* Patients taking medications that may interact with sulfamethoxazole/trimethoprim will be excluded from the study
* Patients taking other probiotics will be excluded from the study
* Patients already taking prophylactic antibiotics will be excluded from the study

Ages: 3 Months to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the rates of bacteriuria among the subjects and the comparison of the two arms. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David R. Roth, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States